CLINICAL TRIAL: NCT00254865
Title: A Comparative Pharmacokinetic Study of EVRA and CILEST in Healthy Female Volunteers
Brief Title: A Comparative Pharmacokinetic Study of ORTHO EVRA (a Transdermal Contraceptive Patch) and CILEST (an Oral Contraceptive) in Healthy Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR003007
Record Dates: First submitted 2005-11-15; First posted 2005-11-17 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-01

CONDITIONS: Contraception; Female Contraception
Keywords: Transdermal contraception; contraceptive; hormonal, steroid contraception; ethinyl estradiol; progesterone; EVRA; CILEST
MeSH Terms: interventions — norelgestromin; Ethinyl Estradiol

INTERVENTIONS:
Drug: EVRA® transdermal contraceptive patch containing 6 mg of norelgestromin and 0.75 mg of ethinyl estradiol (versus CILEST® tablets).

SUMMARY:
The objective of this study is to compare the levels of the hormones norelgestromin, norgestrel, and ethinyl estradiol in the bloodstream of healthy female volunteers administered ORTHO EVRAÂ® (a transdermal contraceptive patch) and CILESTÂ® (an oral contraceptive). The open-label treatment phase of the study consists of two 28-day cycles of one treatment, a washout period of 28 days, and crossover to two 28-day cycles of the other treatment.

DETAILED DESCRIPTION:
ORTHO EVRA® is a combination, monophasic transdermal contraceptive patch containing 6 mg of norelgestromin (NGMN) and 0.75 mg of ethinyl estradiol (EE), and delivering to the systemic circulation an average of 150 µg/day of NGMN and 20 µg/day of EE. CILEST® is an oral contraceptive tablet containing 250 µg of norgestimate (NGM) and 35 µg of ethinyl estradiol (EE). Although the multiple-dose pharmacokinetics of the active serum progestin and estrogen analytes following administration of the ORTHO EVRA® formulation and OrthoCyclen (same as CILEST®) has been evaluated previously in separate studies, the multiple dose pharmacokinetics has not been evaluated in a comparative manner in a single study. The present study is designed to directly compare the total exposure and pharmacokinetics, over comparable time intervals (Week 1 of Cycle 1 and Week 3 of Cycle 2), of NGMN, NG, and EE from ORTHO EVRA® and CILEST® in a single study, designed as a randomized, crossover study. Since EVRA® is worn for 7 days and CILEST® is a once-daily tablet, pharmacokinetics will be estimated over different time periods ORTHO EVRA® (7 days) and CILEST® (Days 1 and/or 7 of a 7 day period) during each cycle. Pharmacodynamic parameters of estrogenicity are determined and compared to assist in the interpretation of the pharmacokinetic data.

This is a single center, randomized, open-label, two-way crossover, pharmacokinetic study of ORTHO EVRA® and CILEST®. The subject population is to be comprised of 32 healthy female volunteers between the ages of 18 and 48 years and having a body mass index (BMI) between 18.0 and 29.9 kg per meter squared. The study consists of a pretreatment phase (a screening period up to 21 days), an open-label treatment phase (two 28-day cycles of 1 treatment, a washout period of 28 days, and cross-over to two 28-day cycles of the other treatment), and a post-treatment phase (a follow-up or early withdrawal visit). Treatment Day 1 is the first day of menses, or within 5 days after the first day of menses. In one treatment period, subjects wear an ORTHO EVRA® patch on their abdomen or buttock (based on the randomization schedule) applied once weekly for 3 consecutive weeks during each of two 28-day cycles. ORTHO EVRA® will be applied and removed by the investigator (or designated study personnel), on Days 1 (application only), 8, 15, and 22 (removal only) of each cycle. In the other treatment period, subjects take CILEST® tablets once daily for the first 21 days of each cycle for two 28-day cycles. CILEST tablets will be administered to the subject with 225 mL (7.5 oz) of water by the investigator or designated personnel on Days 1 through 8 of Cycle 1 and Days 18 through 21 of Cycle 2. On days when the subject is not required to be at the study unit, the subject will self-dose at home (on Days 9 through 21 of Cycle 1 and Days 1 through 17 of Cycle 2). Neither the ORTHO EVRA® patch nor CILEST® tablets are used on Days 22 to 28 (the 4th week) of any cycle, during which subjects may experience withdrawal bleeding. The total duration of the open-label treatment phase is approximately 5 months.

The primary outcome of the study is a comparison of the total exposure and pharmacokinetics, based on comparable intervals, of NGMN, NG, and EE. Blood samples will be drawn during Week 1 of Cycle 1 and Week 3 of Cycle 2 for analysis of plasma NGMN (total and anti and syn isomers), NG, and EE concentrations. Pharmacokinetic parameters, such as Cmax, tmax, and AUC will be estimated by non-compartmental methods. Safety is assessed by monitoring for the incidence and severity of adverse event reports, clinical laboratory tests, vital signs, physical and gynecological examination and an electrocardiogram (ECG). The expectation is that the ratios of exposure between these products and of the ratios of NG/NGMN between these products will be similar. However, the confidence intervals around these ratios are not required to fall within 80-125%. Treatment 1: ORTHO EVRA® transdermal patch, applied once weekly for 3 consecutive weeks of each cycle for two 28-day cycles. Treatment 2: CILEST® tablets, taken once daily by mouth for 21 consecutive days of each cycle, for two 28-day cycles. There is a 28-day washout between treatments.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are not pregnant (as demonstrated by pregnancy tests at screening and admission) or breast feeding, and who have completed their last term pregnancy at least 60 days before the admission visit
* confirmed to be in good health as determined by medical history, physical examination (including vital signs), gynecologic examination (including breast and pelvic exam), laboratory test results, and the absence of evidence of cervical dysplasia (as documented by a Pap smear within 6 months before dosing)
* have a history of regular menstrual cycles, weigh at least 121 pounds (55 kilograms), have a body mass index (BMI) between 18.0 and 29.9 kg per meter squared, and a hematocrit of at least 36%
* are nonsmokers and have not used any tobacco products for at least 6 months before study admission
* Agree not to use any prescription or nonprescription medications for the duration of the study, and if not surgically sterile, agree to use spermicide and barrier contraception, or a nonsteroid-containing intrauterine device as a method of contraception during participation in the study

Exclusion Criteria:

* Subjects with a history or presence of disorders commonly accepted as contraindications to sex hormonal therapy including, but not limited to: deep vein thrombophlebitis or thromboembolic disorders, cerebral vascular or coronary artery disease, chronic untreated hypertension or migraines, benign or malignant liver tumor which developed during the use of oral contraceptives or other estrogen-containing products, or known or suspected estrogen-dependent neoplasia
* presence of disorders commonly accepted as a contraindication to combined oral contraceptive therapy including, but not limited to: undiagnosed abnormal vaginal bleeding, any neurovascular lesion of the eye or serious visual disturbance, any impairment of liver function or liver disease, or kidney disease
* recent history (within 12 months before the admission visit) of alcohol or other substance abuse
* has used steroid-hormonal therapy within 30 days before study admission, received a Depo Provera® injection within 6 months of study admission, currently has Norplant® in place, or has had removal of Norplant within the 60 days before study admission, has used a steroid hormone-containing intra-uterine device (IUD) within 3 months before study admission
* has elevated blood pressure (sitting systolic BP >140 mm Hg or diastolic BP >90 mm Hg)
* has a history or presence of hypersensitivity in response to topical applications (bandages, surgical tape, etc.) or has active inflammation of the skin (dermatitis) or other skin conditions (dermatoses).

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2002-08; Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
A comparison of the total exposure and pharmacokinetics, over comparable time intervals (Week 1 of Cycle 1 and Week 3 of Cycle 2), of NGMN, NG, and EE for ORTHO EVRA® and CILEST®.

SECONDARY OUTCOMES:
Pharmacodynamic measurements [sex hormone-binding globulin (SHBG), corticosteroid binding globulin (CBG), and corticosteroid-binding globulin binding capacity (CBG-BC)] during pre-treatment, Cycle 1, Washout and Cycle 2.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A comparative pharmacokinetic study of EVRA� (a transdermal contraceptive patch) and CILEST� (an oral contraceptive) in healthy female volunteers — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=502&filename=CR003007_CSR.pdf